CLINICAL TRIAL: NCT00082875
Title: A Phase 2 Study of EMD 121974 (Cilengitide, NSC 707544) in Patients With Metastatic Melanoma
Brief Title: Cilengitide in Treating Patients With Unresectable or Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02884; 2003-0988; 6387; N01CM62202 (NIH)
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Stage III Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cilengitide

ARMS (2):
- Arm I (Experimental): Patients receive cilengitide IV over 1 hour on days 1, 4, 8, 11*, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  NOTE: *For the first course only, treatment is omitted on day 11
  Interventions: Drug: cilengitide; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive cilengitide as in arm I at a higher dose.
  Interventions: Drug: cilengitide; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cilengitide — Given IV
  Other Names: EMD 121974
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well cilengitide works in treating patients with unresectable stage III or stage IV melanoma. Cilengitide may stop the growth of melanoma by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the clinical efficacy of EMD 121974 at two different doses in patients with metastatic melanoma by determining the progression-free survival rate at 8 weeks.

SECONDARY OBJECTIVES:

I. To determine the response rate of EMD 121974 in patients with metastatic melanoma.

II. To determine the overall survival in patients who receive EMD 121974. III. To determine the safety and toxicity of EMD 121974 in patients with metastatic melanoma.

IV. To determine the population pharmacokinetics of EMD 121974. V. To determine the biological activity of EMD 121974 in melanoma cells of patients who are treated with the drug.

VI. To evaluate the use of optical imaging and functional dynamic imaging scans in assessing biological activity of EMD 121974.

OUTLINE: This is a randomized, double-blind study. Patients are stratified according to prior systemic treatment (yes vs no), visceral metastases (yes vs no), serum lactic dehydrogenase level (normal vs abnormal), and tumor integrin α_vβ_3 overexpression (yes vs no). Patients are randomized into 1 of 2 treatment arms.

ARM I: Patients receive cilengitide IV over 1 hour on days 1, 4, 8, 11*, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *For the first course only, treatment is omitted on day 11.

ARM II: Patients receive cilengitide as in arm I at a higher dose.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IV or unresectable stage III metastatic melanoma of cutaneous, mucosal or unknown origin
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 15 mm with conventional techniques or with spiral CT scan; in case of obviously visible cutaneous metastatic lesions, the margins of the lesions should be clearly defined and measured in at least one dimension as >= 10 mm
* Patient may have received prior interferon therapy (only in an adjuvant setting for resected stage III melanoma) and/or up to 1 prior systemic treatment regimen (chemotherapy, biotherapy, or biochemotherapy) for stage IV disease; active vaccine therapy will not be considered as "prior systemic treatment"
* Radiographic studies used to assess disease must have been performed within 21 days prior to registration; if a target lesion has been previously embolized, perfused or irradiated, there must be objective evidence of progression before start of therapy to be considered for response assessment
* ECOG performance status ≤ 2 (or Karnofsky ≥ 60%)
* Leukocytes >= 3,000/microL
* Absolute neutrophil count >= 1,500/microL
* Platelets >= 100,000/microL
* Total bilirubin =< 1.5 X institutional upper limit of normal
* ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine =< 1.5 X institutional upper limit of normal
* Patient must have a hemoglobin >= 9 gm/dL (this may be achieved by transfusion if needed) obtained within 14 days prior to registration; in case that PRBC transfusion is needed to obtain a hemoglobin level of >= 9 gm/dL, the hemoglobin level should not be reduced more than 1 gm/dL for at least 1 week
* The effects of EMD 121974 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because antiangiogenic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with metastatic melanoma of choroidal origin
* Patients must not have received the following drugs prior to enrollment: endostatin, angiostatin, bevacizumab or any integrin-targeted drugs
* Subjects who require concurrent treatment with a non-permitted medication (such as anticoagulant therapy other than for flushing of intravenous port device, or used for thrombosis prophylaxis)
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered to grade 1 toxicity from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; however, the following is the exception; patients who have no radiographical evidence of recurrences in the brain for at least 3 months after the complete resection of the brain metastases or who have asymptomatic brain metastases stable for at least 3 months since the whole brain radiation therapy and/or stereotactic radiosurgery will be eligible for this study; patients must not require a steroid treatment for brain metastases
* Subjects with a history of wound-healing disorders, advanced coronary disease (such as unstable angina pectoris or arrhythmia LOWN IV [defined as 2 or more consecutive ventricular premature complexes], cardiac or cardiovascular abnormalities NYHA III/IV), or with a recent history (within 6 months) of peptic ulcer disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because EMD 121974 is an antiangiogenic agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with EMD 121974, breastfeeding should be discontinued if the mother is treated with EMD 121974; lactating women must not breastfeed
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-03; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
PFS | At 8 weeks
  Each dose of EMD 121974 will be analyzed separately.

SECONDARY OUTCOMES:
Response rate, calculated by the ratio of the number of (CR + PR) / total number of treated patients | Up to 4 years
PFS | Up to 4 years
  For each dose of EMD 121974, Kaplan-Meier life table methods and Cox proportional hazards regression modeling will be utilized to analyze progression-free survival.
Overall survival | Up to 4 years
  For each dose of EMD 121974, Kaplan-Meier life table methods and Cox proportional hazards regression modeling will be utilized to analyze overall survival.
Incidence of adverse events graded according to CTCAE version 3.0 | Up to 4 years
  Adverse events will be tabulated by dose of EMD 121974 and toxicity grade.
Population Pharmacokinetics of EMD 121974, including Cmax, tmax, AUClast, t1/2, AUCinf, CL, Vz | Before and 2, 4, and 24 hours after dose of the first dose of courses 1 and 2 and before and 4 hours after dose of the third dose of courses 1 and 2
  Mean and SD will be estimated for each parameter except for tmax, where the median and range will be reported. Plasma concentrations and pharmacokinetic parameters for each dose will be summarized using descriptive statistics and the mean plasma concentrations for each dose will be plotted versus time. Pharmacokinetic parameters will be compared among doses using graphical and statistical analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kim, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States